CLINICAL TRIAL: NCT01514370
Title: ProspeCtive Study to Evaluate Efficacy, Safety and tOlerability of Dietary supplemeNT of Curcumin (BCM95) in Subjects With Active Relapsing MultIple Sclerosis Treated With subcutaNeous Interferon Beta 1a 44 mcg Three Times a Week (TIW)
Brief Title: Dietary Supplement of Curcumin in Subjects With Active Relapsing Multiple Sclerosis Treated With Subcutaneous Interferon Beta 1a
Acronym: CONTAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.P.A., Italy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMR200136-549
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing; Interferon beta 1a; Curcumin
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — Interferon beta-1a; Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- IFN beta 1a 44 mcg TIW + curcumin (BCM95) (Experimental)
  Interventions: Drug: IFN beta 1a 44 mcg TIW; Drug: Curcumin
- IFN beta 1a 44 mcg TIW + placebo (Placebo Comparator)
  Interventions: Drug: IFN beta 1a 44 mcg TIW; Drug: Placebo

INTERVENTIONS:
Drug: IFN beta 1a 44 mcg TIW — Subjects received IFN beta 1a 44 microgram (mcg) subcutaneously TIW for 24 months.
  Other Names: Interferon beta 1a
Drug: Curcumin — Subjects received 500 milligram (mg) curcumin orally twice a day for 24 months.
  Other Names: Rebif; BCM95
  Arms: IFN beta 1a 44 mcg TIW + curcumin (BCM95)
Drug: Placebo — Subjects received placebo matched to curcumin orally twice a day for 24 months.
  Arms: IFN beta 1a 44 mcg TIW + placebo

SUMMARY:
This is a prospective, monocentric, double blind, placebo controlled, two arm study.

Curcumin is derived from the rhizomes of the plant Curcuma longa (common name, turmeric) belonging to the Zingiberaceae family found in South Asian countries, especially India which is the largest producer. BCM95 (bioCurcumin) is a combination of a Curcumin extract and oil to enhance the bio-absorbability in humans. BCM95 may enhance and prolong the antioxidant and anti-inflammatory effects of the standard therapy maintaining a good safety profile.

DETAILED DESCRIPTION:
The subjects must experience at least one Gadolinium (GD) enhancing Magnetic Resonance Imaging (MRI) lesion at the baseline visit or one Multiple Sclerosis (MS) relapse in the last 6 months before the screening visit.

Randomization, in a 1:1 ratio, will be done with two arms:

40 subjects with Interferon (IFN) beta 1 a 44 mcg TIW + Curcumin (BCM 95) and 40 subjects with IFN beta-1a 44 mcg TIW + placebo.

The study will last 42 months: 18 months of enrolment and 24 months of treatment period.

The study consists of 6 visits per subject: screening visit (Visit 0), baseline (Visit 1), a visit 3 months after baseline (Visit 2), 6 months after baseline (Visit 3), 12 months after baseline (Visit 4) and 24 months after baseline (Visit 5).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with early diagnosis (no more than 3 years) of Relapsing Multiple Sclerosis according to the revised McDonald Criteria (2010)
* Subjects currently in treatment with IFN beta-1a 44 mcg TIW, having received this treatment a minimum of 6 months and for not longer than 12 months before enrollment.
* Subjects must experience at least one Gd-enhancing MRI lesion at baseline visit or one MS relapse in the last 6 months before screening visit.
* Males and females between 18 - 60 years of age
* Subjects with Expanded Disability Status Scale (EDSS) between 0-5.5
* No use of oral or systemic corticosteroids or corticotropin (ACTH) within 30 days prior to Screening visit. No use of any Disease Modifying Drug (DMD) (other than IFN beta-1a 44 mcg) 12 months prior to Screening visit
* Be willing and able to comply with the protocol
* Signed informed consent

Exclusion Criteria:

* Pregnancy and breast-feeding
* History of alcohol or drug abuse
* Serious psychiatric disorders
* History or presence of serious or acute gastrointestinal disease such as gastric or duodenal ulcer, ulcerative colitis and inflammatory bowel or Crohn's disease
* Subjects suffering by obstruction of the biliary tract
* Any major medical condition that in the opinion of the Investigator could create a risk to the subject or could affect adherence with the trial protocol.
* Subjects with inadequate haematological function (defined by leukocyte ≤ 2,0 x 10^9 ; platelets ≤ 100 x 10^9; haemoglobin ≤ 12 g/dl for female and ≤ 13 g/dl for male), liver function (defined by AST, ALT, alkaline phosphatase > 2.0 times upper limit of normal), thyroid function (In particular subjects with clinically overt hyperthyroidism or clinically overt hypothyroidism and in any case according to physician's discretion).
* Known hypersensitivity to gadolinium
* Any other condition that would prevent the subject from undergoing an MRI scan (impairment of Kidney function, metal prosthesis etc.)
* Immunosuppressive therapy 12 months before screening visit
* Use of some recognized drugs involved as enzyme substrates, inducers or inhibitors in P450 system
* Use of antiplatelet agents or antihyperlipidemics
* Any contra-indication according to IFN beta 1a 44 mcg Summary of Product Characteristics (SmPC)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono S.P.A., Italy
Locations (1):
- Investigational Site, Naples, Italy

REFERENCES:
- [Derived] Petracca M, Quarantelli M, Moccia M, Vacca G, Satelliti B, D'Ambrosio G, Carotenuto A, Ragucci M, Assogna F, Capacchione A, Lanzillo R, Morra VB. ProspeCtive study to evaluate efficacy, safety and tOlerability of dietary supplemeNT of Curcumin (BCM95) in subjects with Active relapsing MultIple Sclerosis treated with subcutaNeous Interferon beta 1a 44 mcg TIW (CONTAIN): A randomized, controlled trial. Mult Scler Relat Disord. 2021 Nov;56:103274. doi: 10.1016/j.msard.2021.103274. Epub 2021 Sep 21. PMID 34583214

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who had been receiving treatment with subcutaneous interferon (IFN) beta 1a 44 microgram (mcg) three times a week (TIW) for a minimum of 6 months and for not longer than 24 months before enrollment, were enrolled in this study.
Groups:
- IFN Beta 1a 44 mcg TIW + Curcumin (BCM95): Subjects received 500 milligram (mg) curcumin orally twice a day along with IFN beta 1a 44 mcg subcutaneously TIW for approximately 24 months.
- IFN Beta 1a 44 mcg TIW + Placebo: Subjects received placebo matched to curcumin orally twice a day along with IFN beta 1a 44 mcg subcutaneously TIW for approximately 24 months.
Period: Overall Study
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Started | 40 | 40
Safety Population | 38 (The Safety population consisted all randomized subjects who received at least 1 dose of study drug.) | 40 (The Safety population consisted all randomized subjects who received at least 1 dose of study drug.)
Completed | 29 | 24
Not Completed | 11 | 16
Not completed — Protocol Violation | 2 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 3
Not completed — Other | 6 | 7

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (8.6) | 34.3 (9.4) | 35.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 50
  Male | 12 | 18 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Active (New or Enlarging) T2 Lesions Assessed by Magnetic Resonance Imaging (MRI) at Month 12
Description: A single T2 lesion was defined as an area of increased signal on a given 3-millimeters axial image that was not referable to normally hyperintense structures. New T2 lesions were those that appear in areas where on the previous scan no abnormality was detected. All T2 lesions were detected by an MRI scan.
Time Frame: Month 12
Population: ITT population included all randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 40 | 40
Participants | 4 | 7
Statistical Analysis 1: Comparison: IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) vs IFN Beta 1a 44 mcg TIW + Placebo; Test type: Other; p = 0.271, Chi-squared

2. Secondary Outcome: Percentage of Relapse-Free Subjects at Month 12 and Month 24
Description: Relapse was defined as the development of new or the exacerbation of existing neurological symptoms or signs, in the absence of fever, lasting for 24 hours and with a previous period for more than 30 days with a stable or an improving condition.
Time Frame: Month 12 and 24
Population: ITT population included all randomized subjects.
Measure: Number; unit: Percentage of subjects
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 40 | 40
Percentage of subjects
  Month 12 | 75.0 | 67.5
  Month 24 | 60.0 | 50.0

3. Secondary Outcome: Annualized Relapse Rate at Month 12 and 24
Description: Relapse was defined as the development of new or the exacerbation of existing neurological symptoms or signs, in the absence of fever, lasting for 24 hours and with a previous period for more than 30 days with a stable or an improving condition. Annualized relapse rate was calculated by dividing the total number of relapse events by the total number of days subjects participated in the study. This number was then multiplied by 365.25 to get an annualized rate.
Time Frame: Month 12 and 24
Population: ITT population included all randomized subjects. Here, "Number of subjects analyzed" signifies those subjects who were evaluable for this outcome measure. Here "Number analyzed" signifies those subjects who were evaluable for this outcome measure at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Relapse per year
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 12 | 14
Relapse per year
  Month 12: number analyzed (Participants) | 7 | 11
  Month 12 | 1.73 (0.70) | 1.40 (0.65)
  Month 24 | 1.05 (0.73) | 1.14 (0.82)

4. Secondary Outcome: Total Number of Reported Relapses at Month 3, 6, 12 and 24
Description: as for outcome 2
Time Frame: Month 3, 6, 12 and 24
Population: The ITT population included all randomized subjects. Here, "Number of subjects analyzed" signifies those subjects who were evaluable for this outcome measure. Here "Number analyzed" signifies those subjects who were evaluable for this outcome measure at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Relapses
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 7 | 9
Relapses
  Month 3: number analyzed (Participants) | 3 | 5
  Month 3 | 1.00 (0.00) | 1.00 (0.00)
  Month 6: number analyzed (Participants) | 3 | 1
  Month 6 | 1.00 (0.00) | 1.00 (NA) — Standard Deviation could not be estimated as there was only 1 subject analyzed for this arm at the specified timepoint.
  Month 12: number analyzed (Participants) | 4 | 9
  Month 12 | 1.50 (0.58) | 1.00 (0.00)
  Month 24: number analyzed (Participants) | 7 | 4
  Month 24 | 1.57 (0.79) | 1.75 (0.96)

5. Secondary Outcome: Percentage of Subjects Treated With Glucocorticoids Due to Relapses During 24 Months
Description: Relapse was defined as the development of new or the exacerbation of existing neurological symptoms or signs, in the absence of fever, lasting for 24 hours and with a previous period for more than 30 days with a stable or an improving condition. Percentage of subjects treated with glucocorticoids due to relapses during 24 Months were reported here.
Time Frame: Baseline up to Month 24
Population: ITT population included all randomized subjects.
Measure: Number; unit: Percentage of Subjects
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 40 | 40
Percentage of Subjects | 30.0 | 35.0

6. Secondary Outcome: Percentage of Subjects Free From Expanded Disability Status Scale (EDSS) Progression at Month 12 and 24
Description: Disability progression was assessed using EDSS. EDSS is based on a standardized neurological exam and focuses on symptoms that commonly occur in multiple sclerosis (MS) . Overall scores ranges from 0.0 (normal) to 10.0 (death due to MS). Disability progression was defined as an increase of EDSS score of at least 1.0 point compared to baseline for subjects with an EDSS =< 4.0. For subjects with an EDSS= 0 at baseline, EDSS progression was defined as an increase of EDSS score of at least 1.5 point. Percentage of subjects free from EDSS progression at Month 12 and 24 were reported
Time Frame: Month 12 and 24
Population: ITT population included all randomized subjects.
Measure: Number; unit: Percentage of subjects
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 40 | 40
Percentage of subjects
  Month 12 | 92.5 | 82.5
  Month 24 | 90.0 | 85.0

7. Secondary Outcome: Hazard Ratio for Time to First Sustained Expanded Disability Status Scale (EDSS) Progression
Description: EDSS progression is based on a standardized neurological exam and focuses on symptoms that commonly occur in MS. Overall scores ranges from 0.0 (normal) to 10.0 (death due to MS). A sustained progression on EDSS score was defined as an EDSS progression confirmed into two consecutive assessment. EDSS values obtained during clinical attacks are not excluded for the assessment of EDSS progression. However, EDSS values obtained during MS attacks that are not confirmed after two consecutive assessments will be excluded from statistical analysis of confirmed EDSS progression. Hazard ratio for time to first sustained EDSS progression was planned to be reported as per SAP.
Time Frame: Baseline to date at which the first confirmed EDSS progression occurs, assessed up to 24 months
Population: ITT population included all randomized subjects. Here, "Number of subjects analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Ratio
Groups:
- IFN Beta 1a 44 mcg TIW + [Curcumin (BCM95) and Placebo]: Subjects received 500 milligram (mg) curcumin or placebo matched to curcumin orally twice a day along with IFN beta 1a 44 mcg subcutaneously TIW for 24 months.
Arm/Group | IFN Beta 1a 44 mcg TIW + [Curcumin (BCM95) and Placebo]
Number analyzed (Participants) | 79
Ratio | 0.309 [0.023 to 4.115]

8. Secondary Outcome: Percentage of Subjects With Active (New/Enlarging) T2 Lesions at Month 24
Description: as for outcome 1
Time Frame: Month 24
Population: ITT population included all randomized subjects.
Measure: Number; unit: Percentage of subjects
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 40 | 40
Percentage of subjects | 20.0 | 17.5

9. Secondary Outcome: Percentage of Subjects With Combined Unique Active (CUA) Lesions at Month 12 and 24
Description: CUA lesion was defined as new gadolinium (Gd)-enhancing lesions on T1-weighted, or new or enlarging lesions on T2-weighted MRI scans, without double counting.
Time Frame: Month 12 and 24
Population: ITT population included all randomized subjects.
Measure: Number; unit: Percentage of Subjects
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 40 | 40
Percentage of Subjects
  Month 12 | 7.5 | 17.5
  Month 24 | 15.0 | 12.5

10. Secondary Outcome: Mean Number of New Gadolinium (Gd)-Enhancing Lesions at Month 12 and 24
Description: New Gd-enhancing Lesions are a measure of inflammatory activity and were assessed using the Magnetic Resonance Imaging (MRI) scan.
Time Frame: Month 12 and 24
Population: The ITT population included all randomized subjects. Here "Number analyzed" signifies those subjects who were evaluable for this outcome measure at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 40 | 40
Lesions
  Month 12: number analyzed (Participants) | 27 | 26
  Month 12 | 0.19 (0.79) | 0.46 (1.61)
  Month 24: number analyzed (Participants) | 28 | 23
  Month 24 | 0.21 (0.63) | 0.13 (0.63)

11. Secondary Outcome: Mean Number of New T1 (Hypointense) Lesions at Month 12 and 24
Description: Mean number of new T1 (Hypointense) Lesions represents a measure of accumulation of inflammatory disease burden assessed on magnetic resonance imaging (MRI) scans.
Time Frame: Month 12 and 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 40 | 40
Lesions
  Month 12: number analyzed (Participants) | 27 | 25
  Month 12 | 0.52 (1.28) | 0.48 (1.87)
  Month 24: number analyzed (Participants) | 27 | 23
  Month 24 | 0.19 (0.68) | 0.04 (0.21)

12. Secondary Outcome: Cumulative Number of New T1 (Hypointense) Lesions
Description: Cumulative number of new T1 (Hypointense) lesions were reported.
Time Frame: Baseline up to Month 24
Population: The Intent-to-Treat (ITT) population included all randomized subjects. Here "Number of subjects analyzed" included the subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 33 | 33
Lesions | 0.58 (1.32) | 0.39 (1.64)

13. Secondary Outcome: Median Change From Baseline in Whole Brain Volume at Month 12 and 24
Description: Brain tissue volumes are inter-related and represent a measure of neurodegenerative aspects of the disease.
Time Frame: Baseline, Month 12 and 24
Population: As per change in Statistical Analysis Plan, data was not collected for this endpoint
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Median Change From Baseline in Regional Brain Volume at Month 12 and 24
Description: Brain tissue volumes are inter-related and represent a measure of neurodegenerative aspects of the disease.
Time Frame: Baseline, Month 12 and 24
Population: As per change in Statistical Analysis Plan, data was not collected for this endpoint
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Flu-like Symptoms (FLS) Assessed by FLS Scale Score
Description: Flu-like symptoms were measured using FLS score in which subjects were scored as per the presence and intensity of muscle aches, chills, and weakness, each separately, on a scale of 0-3 as follows: 0 = absent; 1 = mild, do not interfere with daily activities; 2 = moderate, sufficient to interfere with daily activities; and 3 = severe, bed rest require. Body temperature also was also recorded to determine the presence of fever using the following scale: 0 (≤ 37.2 °C); 1 (≥ 37.3 °C but < 37.8 °C); 2 (≥ 37.8 but < 38.4 °C); and 3 (≥ 38.4 °C).The scores for each symptom (muscle aches, chills, weakness, body temperature) was added together to provide the combined flu-like symptom score ranging from 0 to 12 where 0 indicates absence of any symptom and 12 indicates the worst severity of the symptoms.
Time Frame: Screening, Baseline, Month 3, 6, 12 and 24
Population: The Safety population included all subjects who received at least one administration of study medication. Here "Number analyzed" signifies those subjects who were evaluable for this outcome measure at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 38 | 40
Units on a scale
  Screening | 2.39 (2.48) | 2.43 (2.34)
  Baseline: number analyzed (Participants) | 16 | 13
  Baseline | 2.22 (2.76) | 2.06 (2.21)
  Month 3: number analyzed (Participants) | 27 | 30
  Month 3 | 1.91 (1.89) | 1.89 (1.74)
  Month 6: number analyzed (Participants) | 27 | 25
  Month 6 | 1.96 (1.83) | 1.91 (2.42)
  Month 12: number analyzed (Participants) | 23 | 24
  Month 12 | 1.45 (1.68) | 1.36 (1.29)
  Month 24: number analyzed (Participants) | 16 | 11
  Month 24 | 1.68 (1.71) | 0.93 (0.92)

16. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Event (TEAE), Serious AE (SAE), TEAE Leading to Death and Discontinuation
Description: AE was defined as any untoward medical occurrence which does not necessarily have a causal relationship with the study drug. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug and up to 24 months. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Month 24
Population: The Safety population included all subjects who received at least one administration of study medication.
Measure: Number; unit: Subjects
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 38 | 40
Subjects
  Subjects with TEAE | 16 | 16
  Subjects with TE-SAE | 1 | 0
  Subjects with TEAEs leading to discontinuation | 1 | 3
  Subjects with TEAEs leading to death | 0 | 0

17. Secondary Outcome: Number of Subjects With Clinical Significant Abnormality in Laboratory Parameters
Description: Laboratory assessment included haematology, chemistry, and urinalysis. Clinical significance was determined by the investigator.
Time Frame: From screening up to Month 24
Population: The Safety population included all subjects who received at least one administration of study medication.
Measure: Number; unit: Subjects
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 38 | 40
Subjects | 9 | 4

18. Secondary Outcome: Number of Subjects With One Concomitant Medication From Baseline up to Month 24
Description: Number of subjects with at least one concomitant medication from baseline up to month 24 were reported.
Time Frame: Baseline up to Month 24
Population: The ITT population included all randomized subjects.
Measure: Number; unit: Subjects
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 40 | 40
Subjects | 28 | 20

19. Secondary Outcome: Time on Treatment (Adherence to Treatment)
Description: Time up to which subjects were adhered to the treatment was reported.
Time Frame: Baseline up to 2.2 years
Population: The Safety population included all subjects who received at least one administration of study medication.
Measure: Median (Full Range); unit: Years
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 38 | 40
Years | 1.93 (0.49) [0.3 to 2.1] | 1.92 (0.60) [0.1 to 2.2]

20. Secondary Outcome: Number of Subjects With Premature Termination From Treatment
Description: Number of subjects with premature termination from treatment were reported.
Time Frame: Baseline up to Month 24
Population: The Intent-to-Treat (ITT) population included all randomized subjects.
Measure: Number; unit: Subjects
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Number analyzed (Participants) | 40 | 40
Subjects
  Adverse event | 1 | 3
  Consent withdrawn | 2 | 1
  Lost to follow up | 0 | 2
  Protocol Violation | 2 | 3
  Unspecified | 6 | 7

21. Secondary Outcome: Hazard Ratio for Time to First Documented Relapse
Description: Relapse was defined as the development of new or the exacerbation of existing neurological symptoms or signs, in the absence of fever, lasting for 24 hours and with a previous period for more than 30 days with a stable or an improving condition. Hazard ratio for time to first documented relapse was planned to be reported as per SAP.
Time Frame: Baseline up to Date at which first Relapse Occurs assessed up to 24 months
Population: ITT population included all randomized subjects.
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | IFN Beta 1a 44 mcg TIW + [Curcumin (BCM95) and Placebo]
Number analyzed (Participants) | 80
Ratio | 0.808 [0.311 to 2.099]

ADVERSE EVENTS:
Time Frame: Baseline up to Month 24
Description: Adverse events were assessed for the safety population. The Safety population included all randomized subjects who received at least 1 administration of study medication.
Arm/Group | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) | IFN Beta 1a 44 mcg TIW + Placebo
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/40
Other Adverse Events (participants affected / at risk) | 16/38 | 16/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) (N=38) | IFN Beta 1a 44 mcg TIW + Placebo (N=40)
Eye abscess (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IFN Beta 1a 44 mcg TIW + Curcumin (BCM95) (N=38) | IFN Beta 1a 44 mcg TIW + Placebo (N=40)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Scotoma (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Venous injury (Injury, poisoning and procedural complications) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 2
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 3 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Astringent therapy (Surgical and medical procedures) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days